CLINICAL TRIAL: NCT04350970
Title: Acute Effects of High-flow Nasal Cannula and Non-invasive Ventilation on Constant-load Exercise Tolerance in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: High-flow Nasal Cannula and Exercise Tolerance in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcelo Alcantara Holanda (Other)
Responsible Party: Sponsor-Investigator, Marcelo Alcantara Holanda, Clinical Investigator, Universidade Federal do Ceara
Organization: Universidade Federal do Ceara (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3.009.159
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: COPD; Rehabilitation; Exercise
Keywords: COPD; High flow nasal therapy; Non-invasive ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: One single COPD group performed 3 differents tests, Control exercise, VNI exercise and HFNT exercise on different days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): The cardiopulmonary exercise test was performed with patient breathing room air.
  Interventions: Other: Control
- NIV (Active Comparator): The cardiopulmonary exercise test was performed with non-invasive ventilation during the test.
  Interventions: Other: Non-invasive ventilation
- HFNT (Active Comparator): The cardiopulmonary exercise test was performed with a High flow nasal therapy during the test.
  Interventions: Other: High flow nasal therapy

INTERVENTIONS:
Other: High flow nasal therapy — All patients underwent two cardiopulmonary exercises with constant-load at 90% of the peak workload. The high flow nasal therapy was used during all exercise test.
  Arms: HFNT
Other: Non-invasive ventilation — All patients underwent two cardiopulmonary exercises with constant-load at 90% of the peak workload. The NIV was used during all exercise test.
  Arms: NIV
Other: Control — All patients underwent two cardiopulmonary exercises with constant-load at 90% of the peak workload. The control test was performed with no additional therapy.
  Arms: Control

SUMMARY:
Patients with COPD are often unable to sustain a sufficient workload during exercise. The use of external strategies to improve exercise tolerance, such as non-invasive ventilation (NIV) and high-flow nasal therapy (HFNT) have been used. The objective was to evaluate and compare the acute effects of HFNT and NIV during exercise on cardiorespiratory parameters, dyspnea, exercise tolerance and comfort in patients with moderate to severe COPD.

DETAILED DESCRIPTION:
The patients underwent an initial clinical examination, with anthropometric evaluation, blood gas analysis, pulmonary function tests and measurement of maximum respiratory pressures. The exercise protocol started in the sector of Ergometry and Cardiopulmonary Exercise Testing. After completing the maximum incremental cardiopulmonary exercise test, two additional visits were scheduled for the three constant load tests. All patients studied underwent an evaluation of cardiopulmonary exercise testing (CPET). During maximum-incremental CPET, breath by breath: oxygen consumption (V̇O2, mL/min), carbon dioxide production (V̇CO2, mL/min), respiratory exchange rate (RER), minute ventilation VE (L/min), respiratory rate (bpm), equivalent ventilation for O2 and CO2 (V̇E/V̇O2 and V̇E/V̇CO2). In addition, cardiac monitoring was performed by 12-lead electrocardiogram (ECG) throughout the procedure. On the day of the experiment, the patients underwent two cardiopulmonary exercises with constant-load at 90% of the previously determined peak, separated by an interval of at least 1 hour.

The NIV parameters were adjusted for each patient with Trilogy 100 (Philips™). Spontaneous ventilation mode was set before the protocol for all patients, and a previous period of NIV adaptation was performed to titrate the inspiratory and expiratory pressures. The adaptation period started with the minimum Inspiratory Positive Airway Pressure (IPAP) value of 15cmH2O, and, every 2 minutes, increasing the pressure every 2 cmH2O according to the patient's tolerance.16 The Expiratory Positive Airway Pressure (EPAP) was programmed to vary between 4 and 6 cmH2O. Before the start of the examination, an adaptation was performed with the selected mask and initial ventilator settings for 20 min. No additional oxygen was offered.

The high flow system used was Optiflow® (Fisher & Paykel Healthcare, Auckland, New Zealand). Before the test, flow titration was performed for the patient, which started with the administration of a minimum gas flow of 30L/min and, every 2 minutes, the flow was increased by 5L/min according to patient tolerance. The test only started after 20 minutes of adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Previous COPD
* FEV1 ≤ 50%
* Optimized medication

Exclusion Criteria:

* COPD Exacerbation
* Cardiac disease
* Previous neurologic disorders
* Unable to complete all protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Exercise dinamic hyperinflation | one week after all tests
  To determine the dinamic hyperinflation during exercise test with 3-different situations , Control, NIV and HFNT. During all testes the dinamic hyperinflation will be measured by inspiratory capacity (at rest and at the end o exercise test) and will be demonstrated as porcentage os maximum.
Exercise Tolerance | one week after all tests
  To determine the exercise tolerance with 3-different situations , Control, NIV and HFNT. Time of exercise test will be measured to determine which test could be the best for COPD patients. In additional, the workload will (treadmill inclination and speed) be check to show which intervention has the better response.

SECONDARY OUTCOMES:
Dyspnea | one week after all tests
  To determine the dyspnea during exercise test with 3-different situations , Control, NIV and HFNT. After all situations, Borg scale will be performed to check the dyspnea score at the end of exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No
This is study will be submitted to a medical journal.